CLINICAL TRIAL: NCT05112107
Title: Evaluation Of Strategies For Improving Ketogenic Diet Compliance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Erasmo Barbante Casella, Clinical Professor, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CAAE19812919.2.0000.0068
Record Dates: First submitted 2021-08-15; First posted 2021-11-08 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: Epilepsy; Ketogenic Dieting; Compliance, Treatment
MeSH Terms: conditions — Epilepsy; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention)
- Intervention (Experimental)
  Interventions: Behavioral: Culinary workshops

INTERVENTIONS:
Behavioral: Culinary workshops — Approved ketogenic recipes will be applied in educational cooking workshops at the ketogenic diet clinic at Instituto da Criança HCFMUSP.
  Arms: Intervention

SUMMARY:
In order to increase adherence to ketogenic diet treatment, palatability of meals and diversify the foods offered to patients a ketogenic kitchen will be created. Intervention: Incorporation of culinary workshops and supply of recipes for patients undergoing ketogenic diet treatment at Instituto da Criança - HCFMUSP.

DETAILED DESCRIPTION:
Introduction: The ketogenic diet is a therapeutic option for the control of drug-resistant epileptic seizures. It is based on high fat consumption, protein control and carbohydrate restriction. As a result, the body uses fat as an energy substrate instead of glucose. Changing the patient's daily menu and eating routine is hard and requires dedication from the caregiver for the best therapeutic result. In clinical practice, the diet becomes monotonous and poorly accepted by the patient over time. Besides, there is a difficulty in understanding nutritional guidelines. It is necessary to develop strategies to increase adherence to treatment, palatability of meals and diversify the foods offered to patients. Objective: To evaluate the effectiveness of creating a ketogenic kitchen in improving compliance of patients with CD in the outpatient clinic of Instituto da Criança - HCFMUSP. Methods: this work will be carried out in 4 steps: (1st) Creation and validation of a questionnaire of ketogenic diet compliance, (2nd) Creation of ketogenic recipes of easy preparation and low cost, (3rd) Incorporation of culinary workshops and supply of recipes for patients undergoing treatment at Instituto da Criança - HCFMUSP and (4th) Application of the questionnaire of ketogenic diet compliance.

ELIGIBILITY:
Inclusion Criteria:

* Patients 0 to 18 years old;
* Clinical indication of a classic ketogenic diet;
* Predominantly oral feeding.

Exclusion Criteria:

* Patients using exclusive gastrostomy;
* Patients with other types of KD than Classical KD.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-12-30 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2024-05-05 (Estimated)

PRIMARY OUTCOMES:
Ketogenic diet compliance score | through study completion, an average of 2 years
  Ketogenic diet compliance score will be obtained through a validated questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Erasmo Casella, PhD, Principal Investigator — University of Sao Paulo General Hospital
Locations (1):
- Instituto da Criança Hospital das Clinicas da Universidade de São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No